CLINICAL TRIAL: NCT04658784
Title: Barbed Suture Versus Non-Barbed Suture for Posterior Colporrhaphy: A Randomized Controlled Trial
Brief Title: Barbed Suture Versus Non-Barbed Suture for Posterior Colporrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00082745; #04-20-01 (Other: Atrium)
Record Dates: First submitted 2020-11-19; First posted 2020-12-08 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Rectocele
Keywords: pelvic organ prolapse; barbed suture; posterior colporrhaphy; posterior repair; pain
MeSH Terms: conditions — Rectocele; Pelvic Organ Prolapse; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Receives posterior colporrhaphy closure using standardized technique with 2-0 V-Loc 90TM, Medtronic
  Interventions: Device: 2-0 dioxanone, glycolide and trimethylene carbonate
- Control (Active Comparator): Receives posterior colporrhaphy closure using standardized technique with conventional 2-0 PDS® Ethicon
  Interventions: Device: 2-0 polydioxanone

INTERVENTIONS:
Device: 2-0 dioxanone, glycolide and trimethylene carbonate — delayed absorbable, monofilament barbed suture
  Other Names: 2-0 V-Loc 90TM (Medtronic)
  Arms: Intervention
Device: 2-0 polydioxanone — delayed absorbable, monofilament non-barbed suture
  Other Names: 2-0 PDS® (Ethicon)
  Arms: Control

SUMMARY:
The aim of this randomized clinical trial is to compare barbed suture versus non-barbed suture at the time of posterior repair on postoperative pain scores as measured by a visual analog scale (VAS) at 6 weeks.

Study participants are randomized to use of barbed suture (2-0 V-Loc 90TM, Medtronic) or non-barbed suture (2-0 Polydioxanone, PDS® EthiconTM) in a standardized technique for posterior colporrhaphy at the time of posterior repair.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a growing concern for the aging female population, and symptomatic women often require surgical intervention. Approximately 200,000 surgical procedures for POP are performed annually in the United States. This number is anticipated to increase with the growth in the aging population.1 Surgical prolapse repairs are often categorized into either mesh augmented or native tissue repairs. During a native tissue repair, the surgeon uses a woman's natural tissue to repair the prolapse without augmenting the repair with synthetic mesh.

Women often have post-operative pain with native tissue posterior colporrhaphy. Native tissue posterior repairs are performed to address symptomatic posterior compartment prolapse, defects in the rectovaginal fibromuscularis, and/or a widened genital hiatus. This type of repair may improve obstructed defecatory dysfunction and bulge symptoms, but can be associated with postoperative pelvic pain and dyspareunia. Paraiso et al evaluated three surgical techniques for posterior colporrhaphy (site-specific, midline plication, and porcine graft) and found no difference in overall symptom improvement, quality of life, and post-operative sexual function. Regardless of the technique used, a posterior colporrhaphy can cause considerable postoperative pain and can contribute to de novo dyspareunia in 9-20% of women. Most studies evaluating pain after posterior colporrhaphy tend to focus on various methods of analgesia and surgical technique rather than the suture materials used.

Suture choice may contribute to postoperative pain at the time of posterior colporrhaphy. There are few studies evaluating suture in the posterior compartment with no defined standard suture material for posterior colporrhaphy. Available studies, when comparing subjective bulge and quality of life outcomes, do not demonstrate superiority of one suture type over the other. Delayed absorbable suture has the benefit of retaining tensile strength for approximately 3 months. Delayed absorbable suture material itself, however, can remain in place for up to 8 months. These properties may decrease postoperative pain by decreasing knot burden. Barbed suture has been successfully applied to vaginal cuff closure, myomectomy, sacrocolpopexy mesh attachment, and closure of bowel and bladder injuries with demonstrated reduced operative times. To date, no studies have evaluated the impact of barbed suture on postoperative pain or surgical time after posterior colporrhaphy.

The primary objective for this study is to compare delayed absorbable barbed suture versus non-barbed delayed absorbable suture at the time of posterior repair on post-operative posterior compartment pain scores, as measured by the Visual Analog Scale (VAS), at 6 weeks

Secondary objectives include a comparison of VAS pain scores in the posterior compartment at 6-months, evaluation of operative time for posterior repair in minutes, evaluation of suture burden and pelvic pain on examination of the posterior compartment, evaluation of pain versus the length of a repair, evaluation of postoperative patient quality of life (QoL) using series of standardized questionnaires, evaluation of suture cost, and a comparison of anatomical and surgical failure in the posterior compartment.

Participants will be approached for participation preoperatively. Baseline demographic data will be abstracted from the medical record. A baseline Pelvic Organ Prolapse Quantification (POP-Q) and pelvic myofascial exam will be performed. Baseline VAS and validated questionnaires: Pelvic Floor Distress Inventory-20 (PFDI-20) sub-scales Colorectal-Anal Distress Inventory-8 (CRADI-8) and Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire- 12 (PISQ-12 )will be completed. Participants will be randomized in the operating room after posterior vaginal dissection to either barbed or non-barbed suture in a standardized technique. All concurrent minimally invasive pelvic reconstructive surgical procedures are allowed. Randomization will be stratified for minimally invasive (robotic or laparoscopic) versus vaginal surgery.

Perioperative care is standardized.

Participants will be scheduled for a post-operative follow up visit at approximately 6 weeks. At this visit they will have a structured postoperative interview and pelvic examination, including POP-Q, standardized assessment of suture burden and myofascial trigger points. They will also complete a VAS and validated questionnaires. Participants will be called at approximately 6 months after their original surgery. They will have a structured interview and complete VAS and complete validated questionnaires.

Adverse postoperative outcomes will be collected at each visit.

Investigators will use a standard deviation estimate of 23.4mm to detect a difference on a 100mm VAS for pain. Accounting for a 15% drop-out rate, the investigators aim to enroll 64 participants with 32 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18yo or older
* English speaking
* Planned posterior colporrhaphy with or without perineorrhaphy with concomitant surgical procedures allowed

Exclusion Criteria:

* Documented allergy or contraindication to use of suture material
* Prior mesh in posterior compartment
* Planned colpocleisis
* Current or prior rectovaginal fistula
* Planned sacrospinous ligament fixation procedure
* Chronic pelvic pain diagnosis
* Chronic narcotic medication use
* Active vulvodynia
* Non-English speaking
* Inability to provide informed consent
* Planned combined colorectal/anorectal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study involves women undergoing surgery for pelvic organ prolapse.
Enrollment: 72 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Merriman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones KA, Shepherd JP, Oliphant SS, Wang L, Bunker CH, Lowder JL. Trends in inpatient prolapse procedures in the United States, 1979-2006. Am J Obstet Gynecol. 2010 May;202(5):501.e1-7. doi: 10.1016/j.ajog.2010.01.017. Epub 2010 Mar 11. PMID 20223444
- [Background] Kahn MA, Stanton SL. Posterior colporrhaphy: its effects on bowel and sexual function. Br J Obstet Gynaecol. 1997 Jan;104(1):82-6. doi: 10.1111/j.1471-0528.1997.tb10654.x. PMID 8988702
- [Background] Karjalainen PK, Mattsson NK, Nieminen K, Tolppanen AM, Jalkanen JT. The relationship of defecation symptoms and posterior vaginal wall prolapse in women undergoing pelvic organ prolapse surgery. Am J Obstet Gynecol. 2019 Nov;221(5):480.e1-480.e10. doi: 10.1016/j.ajog.2019.05.027. Epub 2019 May 22. PMID 31128111
- [Background] Paraiso MF, Barber MD, Muir TW, Walters MD. Rectocele repair: a randomized trial of three surgical techniques including graft augmentation. Am J Obstet Gynecol. 2006 Dec;195(6):1762-71. doi: 10.1016/j.ajog.2006.07.026. PMID 17132479
- [Background] Komesu YM, Rogers RG, Kammerer-Doak DN, Barber MD, Olsen AL. Posterior repair and sexual function. Am J Obstet Gynecol. 2007 Jul;197(1):101.e1-6. doi: 10.1016/j.ajog.2007.03.054. PMID 17618777
- [Background] Mowat A, Maher D, Baessler K, Christmann-Schmid C, Haya N, Maher C. Surgery for women with posterior compartment prolapse. Cochrane Database Syst Rev. 2018 Mar 5;3(3):CD012975. doi: 10.1002/14651858.CD012975. PMID 29502352
- [Background] Evans SKL, Abimbola O, Myers EM, Tarr ME. A Novel Injection Technique for Extended-Release Local Anesthetic After Posterior Colporrhaphy and Perineorrhaphy: A Randomized Controlled Study. Female Pelvic Med Reconstr Surg. 2021 Jun 1;27(6):344-350. doi: 10.1097/SPV.0000000000000855. PMID 32384288
- [Background] Luck AM, Galvin SL, Theofrastous JP. Suture erosion and wound dehiscence with permanent versus absorbable suture in reconstructive posterior vaginal surgery. Am J Obstet Gynecol. 2005 May;192(5):1626-9. doi: 10.1016/j.ajog.2004.11.029. PMID 15902168
- [Background] Madhuvrata P, Glazener C, Boachie C, Allahdin S, Bain C. A randomised controlled trial evaluating the use of polyglactin (Vicryl) mesh, polydioxanone (PDS) or polyglactin (Vicryl) sutures for pelvic organ prolapse surgery: outcomes at 2 years. J Obstet Gynaecol. 2011 Jul;31(5):429-35. doi: 10.3109/01443615.2011.576282. PMID 21627429
- [Background] Allahdin S, Glazener C, Bain C. A randomised controlled trial evaluating the use of polyglactin mesh, polydioxanone and polyglactin sutures for pelvic organ prolapse surgery. J Obstet Gynaecol. 2008 May;28(4):427-31. doi: 10.1080/01443610802150077. PMID 18604681
- [Background] Bergman I, Soderberg MW, Kjaeldgaard A, Ek M. Does the choice of suture material matter in anterior and posterior colporrhaphy? Int Urogynecol J. 2016 Sep;27(9):1357-65. doi: 10.1007/s00192-016-2981-0. Epub 2016 Mar 2. PMID 26935306
- [Background] Greenberg JA, Clark RM. Advances in suture material for obstetric and gynecologic surgery. Rev Obstet Gynecol. 2009 Summer;2(3):146-58. PMID 19826572
- [Background] Greenberg JA, Goldman RH. Barbed suture: a review of the technology and clinical uses in obstetrics and gynecology. Rev Obstet Gynecol. 2013;6(3-4):107-15. PMID 24920976
- [Background] Iavazzo C, Mamais I, Gkegkes ID. The Role of Knotless Barbed Suture in Gynecologic Surgery: Systematic Review and Meta-Analysis. Surg Innov. 2015 Oct;22(5):528-39. doi: 10.1177/1553350614554235. Epub 2014 Oct 15. PMID 25320107
- [Background] Chamsy D, King C, Lee T. The use of barbed suture for bladder and bowel repair. J Minim Invasive Gynecol. 2015 May-Jun;22(4):648-52. doi: 10.1016/j.jmig.2015.01.030. Epub 2015 Feb 7. PMID 25659867
- [Background] Wiggins T, Majid MS, Markar SR, Loy J, Agrawal S, Koak Y. Benefits of barbed suture utilisation in gastrointestinal anastomosis: a systematic review and meta-analysis. Ann R Coll Surg Engl. 2020 Feb;102(2):153-159. doi: 10.1308/rcsann.2019.0106. Epub 2019 Sep 11. PMID 31508982
- [Background] Maher CF, Qatawneh AM, Baessler K, Schluter PJ. Midline rectovaginal fascial plication for repair of rectocele and obstructed defecation. Obstet Gynecol. 2004 Oct;104(4):685-9. doi: 10.1097/01.AOG.0000139833.48063.03. PMID 15458886
- [Background] Christmann-Schmid C, Wierenga AP, Frischknecht E, Maher C. A Prospective Observational Study of the Classification of the Perineum and Evaluation of Perineal Repair at the Time of Posterior Colporrhaphy. Female Pelvic Med Reconstr Surg. 2016 Nov/Dec;22(6):453-459. doi: 10.1097/SPV.0000000000000314. PMID 27636214
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Crisp CC, Bandi S, Kleeman SD, Oakley SH, Vaccaro CM, Estanol MV, Fellner AN, Pauls RN. Patient-controlled versus scheduled, nurse-administered analgesia following vaginal reconstructive surgery: a randomized trial. Am J Obstet Gynecol. 2012 Nov;207(5):433.e1-6. doi: 10.1016/j.ajog.2012.06.040. Epub 2012 Jun 20. PMID 22863282
- [Background] Barber MD, Brubaker L, Nygaard I, Wheeler TL 2nd, Schaffer J, Chen Z, Spino C; Pelvic Floor Disorders Network. Defining success after surgery for pelvic organ prolapse. Obstet Gynecol. 2009 Sep;114(3):600-609. doi: 10.1097/AOG.0b013e3181b2b1ae. PMID 19701041
- [Background] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Lee JS, Hobden E, Stiell IG, Wells GA. Clinically important change in the visual analog scale after adequate pain control. Acad Emerg Med. 2003 Oct;10(10):1128-30. doi: 10.1111/j.1553-2712.2003.tb00586.x. PMID 14525749
- [Background] Westermann LB, Crisp CC, Mazloomdoost D, Kleeman SD, Pauls RN. Comparative Perioperative Pain and Recovery in Women Undergoing Vaginal Reconstruction Versus Robotic Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):95-100. doi: 10.1097/SPV.0000000000000368. PMID 28067743
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle T, Warren DK, Lowder JL. Development of a standardized, reproducible screening examination for assessment of pelvic floor myofascial pain. Am J Obstet Gynecol. 2019 Mar;220(3):255.e1-255.e9. doi: 10.1016/j.ajog.2018.11.1106. Epub 2018 Dec 7. PMID 30527941
- [Background] He S, Falk K, Kannan A, Kelley RS. An Alternative Approach to Posterior Colporrhaphy Plication Using Delayed Absorbable Unidirectional Barbed Suture. Female Pelvic Med Reconstr Surg. 2020 Feb;26(2):107-110. doi: 10.1097/SPV.0000000000000828. No abstract available. PMID 31990797
- [Background] Culligan PJ. Surgical repair of the posterior compartment. Clin Obstet Gynecol. 2005 Sep;48(3):704-12. doi: 10.1097/01.grf.0000170426.61066.34. No abstract available. PMID 16012237

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to 6-week Follow-up
Arm/Group | Intervention | Control
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0
Period: 6-month Follow-up
Arm/Group | Intervention | Control
Started | 36 | 36
Completed | 34 | 31
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (10.5) | 58.2 (11.0) | 57.9 (10.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 34 | 68
  Black | 2 | 1 | 3
  Other | 0 | 1 | 1
BMI kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (3.9) | 28.3 (4.9) | 28.0 (4.4)
Tobacco use [Count of Participants; unit: Participants] | 1 | 1 | 2
Sexually active [Count of Participants; unit: Participants] | 22 | 27 | 49
Vaginal estrogen use [Count of Participants; unit: Participants] | 3 | 7 | 10
Total Pelvic Organ Prolapse Quantification (POP-Q) Stage [Count of Participants; unit: Participants] — Pelvic Organ Prolapse-Quatification (POP-Q) Stage 0-IV, where stage 0 is the least severe and equal to no prolapse present and IV most severe stage of prolapse equal to complete vaginal eversion/ uterine procidentia. Total POP-Q stage is the highest stage of any compartment (anterior, posterior, or apical) calculated by using the leading edge as point of measurement.
  Participants
    POP-Q Stage 0 | 0 | 0 | 0
    POP-Q Stage I | 0 | 1 | 1
    POP-Q Stage II | 27 | 16 | 43
    POP-Q Stage III | 8 | 16 | 24
    POP-Q Stage IV | 1 | 3 | 4
Posterior Compartment Pelvic Organ Prolapse Quantification (POP-Q) Stage (0-IV) [Count of Participants; unit: Participants] — Pelvic Organ Prolapse-Quatification (POP-Q) Stage 0-IV, where stage 0 is the least severe and equal to no prolapse present and IV most severe stage of prolapse equal to complete vaginal eversion/ uterine procidentia. Posterior compartment POP-Q stage is calculated using the leading edge of posterior prolapse as the point of measurement.
  Participants
    POP-Q Stage 0 | 2 | 1 | 3
    POP-Q Stage I | 8 | 4 | 12
    POP-Q Stage II | 26 | 25 | 51
    POP-Q Stage III | 0 | 5 | 5
    POP-Q Stage IV | 0 | 1 | 1
Prior pelvic reconstructive surgery [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Posterior Compartment Pain Scores - Posterior Repair
Description: To compare delayed absorbable barbed suture versus non-barbed delayed absorbable suture at the time of posterior repair on post-operative posterior compartment pain scores, as measured by the Visual Analog Scale (VAS).The VAS is a validated scale that is ranges from 0-100mm. 0mm is equivalent to "no pain" and is located on the left. 100mm is equivalent to "worst possible pain" and is located on the right. Reported as categorical variable no pain (VAS 0), low pain (VAS 1-33), moderate pain (VAS 34-66), and high pain (VAS 67-100).
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Participants
  no pain (VAS 0) | 32 | 29
  low pain (VAS 1-33) | 2 | 4
  moderate pain (VAS 34-66) | 1 | 2
  high pain (VAS 67- 100) | 1 | 1
  missing | 0 | 0
Statistical Analysis 1: Comparison: Intervention vs Control; OR calculated from logistic regression model, evaluating mean change in baseline VAS to 6-weeks; Test type: Superiority; p = 0.32, Regression, Logistic — OR, 95% CI, and p-values for outcomes adjusted for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery). P-value for VAS at 6-weeks was not adjusted for multiple comparisons; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.13 to 1.92]

2. Secondary Outcome: Post-operative Posterior Compartment Pain Scores
Description: To compare visual analog scale (VAS) pain scores in the posterior compartment. The VAS is a validated scale that is ranges from 0-100mm. 0mm is equivalent to "no pain" and is located on the left. 100mm is equivalent to "worst possible pain" and is located on the right. Reported as categorical variable no pain, low pain, moderate pain and high pain. Reported as categorical variable no pain (VAS 0), low pain (VAS 1-33), moderate pain (VAS 34-66), and high pain (VAS 67-100).
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Participants
  no pain (VAS 0) | 33 | 26
  low pain (VAS 1-33) | 1 | 1
  moderate pain (VAS 34-66) | 0 | 1
  high pain (VAS 67- 100) | 0 | 0
  missing | 2 | 8
Statistical Analysis 1: Comparison: Intervention vs Control; OR calculated from logistic regression model, evaluating mean change in baseline VAS to 6-weeks; Test type: Superiority; p = 1.0, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.04 to 5.65]

3. Secondary Outcome: Operative Time
Description: To evaluate operative time for posterior repair in minutes.
Time Frame: Time of Surgery
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Minutes
  Total procedure surgical time | 146 [75 to 180] | 168 [114 to 192]
  Posterior repair surgical time | 21 [15.5 to 28.5] | 20.5 [15.5 to 31.5]

4. Secondary Outcome: Suture Burden
Description: To evaluate amount of suture burden present at time of surgery in posterior by compartment by measuring total amount of delayed absorbable suture used for posterior colporrhaphy in centimeters.
Time Frame: At time of surgery (Intraoperative)
Measure: Median (Inter-Quartile Range); unit: centimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
centimeters | 10.5 [7.9 to 14.4] | 26.9 [14.9 to 48.6]

5. Secondary Outcome: Change in Bowel Function Scores
Description: To evaluate change in bowel function using the Pelvic Floor Distress Inventory- 20 (PFDI-20) sub-scale Colorectal-Anal Distress Inventory-8 (CRADI-8). Total score (range 0 to 100) with the higher the score the more distress.
Time Frame: Baseline, Week 6, and month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline | 36.4 (20.8) | 36.6 (19.0)
  6 weeks | 18.1 (14.4) | 18.1 (14.9)
  Change from baseline to 6 weeks | -18.2 (19.6) | -18.6 (22.7)
  6 months | 12.3 (12.7) | 9.6 (12.8)
  Change from baseline to 6 months | -24.1 (22.6) | -27.9 (19.7)
Statistical Analysis 1: Comparison: Intervention vs Control; Differences in mean change and 95% CI generated from general linear models. Change from baseline to 6- weeks; Test type: Superiority; p = 1.0, Regression, Linear — Adjust for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery); Mean Difference (Net) = 2.6, 95% CI 2-sided [-3.5 to 8.7]
Statistical Analysis 2: Comparison: Intervention vs Control; Differences in mean change and 95% CI generated from general linear models. Change from baseline to 6-months; Test type: Superiority; Regression, Linear — Adjust for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery); Mean Difference (Net) = -1.2, 95% CI 2-sided [-5.6 to 3.2]

6. Secondary Outcome: Change in Pelvic Organ Prolapse Symptoms
Description: To evaluate change in pelvic organ prolapse symptoms using the Pelvic Floor Distress Inventory- 20 (PFDI-20) sub-scale the Pelvic Organ Prolapse Distress Inventory- 6 (POPDI-6). Total score (range 0 to 100) with the higher the score the more distress.
Time Frame: Baseline, Week 6, and Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline | 53.4 (19.5) | 52.1 (18.2)
  6 weeks | 13.8 (13.0) | 11.2 (12.9)
  change from baseline to 6 weeks | -39.6 (20.7) | -40.9 (23.4)
  6 months | 7.2 (9.6) | 8.3 (9.0)
  Change from baseline to 6 months | -46.7 (18.8) | -43.1 (20.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Differences in mean change and 95% CI generated from general linear models. Change in baseline to 6-weeks; Test type: Superiority; p = 1.0, Regression, Linear — Adjust for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery); Mean Difference (Net) = 0.2, 95% CI 2-sided [-6.6 to 6.9]
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority — Differences in mean change and 95% CI generated from general linear models. Change in baseline to 6-months; p = 1, Regression, Linear — Adjusted for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery); Mean Difference (Net) = 2.8, 95% CI 2-sided [-3.1 to 8.6]

7. Secondary Outcome: Change in Postoperative Sexual Function Scores
Description: To evaluate postoperative sexual function using the Pelvic Organ Prolapse-Urinary Incontinence Sexual Function Questionnaire (PISQ-12). Total score (range 0 to 48) with a lower score associated with poorer/worse sexual function.
Time Frame: Month 6
Population: Different number of patients were sexually active at measured time points, baseline and 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 22
score on a scale
  Baseline | 28.1 (5.0) | 26.9 (6.3)
  6 months: number analyzed (Participants) | 22 | 16
  6 months | 33.1 (3.2) | 31.7 (4.6)
  Change from baseline to 6 months: number analyzed (Participants) | 15 | 21
  Change from baseline to 6 months | 3.9 (6.8) | 4.6 (4.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Differences in mean change and 95% CI generated from general linear models. Change from baseline to 6 months; Test type: Superiority; p = 1.0, Regression, Linear — Adjusted for baseline value and type of surgery (vaginal or vaginal + minimally invasive surgery); Mean Difference (Net) = -1.6, 95% CI 2-sided [-4.4 to 1.3]

8. Secondary Outcome: Number of Patients With Early Anatomic Recurrence
Description: To evaluate anatomical failure of posterior compartment using a standard definition of anatomical cure will be defined as Ba or Bp at </= 0 on POP-Q examination (i.e.at or beyond hymenal ring)
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Participants | 0 | 0

9. Secondary Outcome: Number of Patients With Subjective Failure
Description: To evaluate subjective failure of posterior compartment using a negative response on POPDI-6 portion of the PFDI-20 questionnaire to questions: "Do you usually have a sensation of bulging or protrusion from the vaginal area?" and "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?"
Time Frame: Week 6 and Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Participants
  6 weeks | 0 | 0
  6 months | 1 | 2

10. Secondary Outcome: American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) 30-day Postoperative Complications.
Description: To evaluate differences in adverse outcomes, using number of adverse events (AEs) as defined by the American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) 30-day postoperative complications criteria. These criteria were reviewed at the week 6 data collection time interval.
Time Frame: 30 days
Population: Comparison of 30 day ACS NSQIP complications in intervention and control groups.
Measure: Number; unit: Adverse events
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 36
Adverse events
  Urinary tract infection (UTI) | 5 | 3
  Surgical site infection (SSI) | 0 | 1
  Readmission | 1 | 0
  Return to the operating room (OR) | 1 | 0
  Unplanned reintubation | 0 | 1

11. Secondary Outcome: Surgery Specific Adverse Events (AEs) Measured at 6-months.
Description: To evaluate differences in adverse outcomes, using number of surgery specific adverse events.
Time Frame: month 6
Population: Analysis of surgery specific adverse events in intervention and control groups.
Measure: Number; unit: Adverse events
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 31
Adverse events
  de novo dyspareunia | 4 | 5
  new or worsening pelvic pain >3months | 1 | 4
  New or worsening constipation > 3 months | 2 | 1
  New fecal incontinence | 1 | 1
  Nerve injury | 1 | 0
  Other | 1 | 0
  Classified as Severe Adverse Event (SAE) | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 6 weeks, 6 months and 12 months time points.
Description: No difference in definitions or collection.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/36
Other Adverse Events (participants affected / at risk) | 14/36 | 13/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=36) | Control (N=36)
Nerve entrapment (Nervous system disorders) | 1 (1) | 1 (1) — A single patient from intervention group was readmitted and returned to the operating room within 30-days of surgery due to severe right sided vaginal pain and concern for nerve entrapment after utter-sacral ligament suspension.
Pelvic pain (Nervous system disorders) | 1 (1) | 1 (1) — Single patient in control group with severe pelvic pain >3 months requiring multiple medical interventions for treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=36) | Control (N=36)
Surgical site infection (Infections and infestations) | 1 (1) | 1 (1) — Not associated with posterior repair.
Urinary tract infection (UTI) (Infections and infestations) | 5 (5) | 3 (3)
New or worsening pelvic pain > 3months (Nervous system disorders) | 1 (1) | 4 (4)
De novo dyspareunia (Reproductive system and breast disorders) | 4 (4) | 5 (5)
New fecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
New or worsening constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Ovarian vein thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04658784/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT04658784/ICF_001.pdf